CLINICAL TRIAL: NCT00285896
Title: The Effect of 48 Hours of GLP-1 Infusion During Long-Time Fasting on Glycaemia and Counterregulatory Hormones
Brief Title: GLP-1 Infusion and Long-Time Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Professor Ole E. Schmitz, University of Aarhus, department of Pharmacology
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004-0172
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2008-07-11 (Estimated); Status verified 2008-07

CONDITIONS: Type 2 Diabetes
Keywords: GLP-1; fasting; hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fasting; Hypoglycemia | interventions — glucagon-like peptide 1 (7-36)amide; Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): GLP-1
  Interventions: Drug: Glucagon-like-peptide-1 (7-36) amide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glucagon-like-peptide-1 (7-36) amide — Continuous, subcutaneous GLP-1 at a dose of 4.8 pmol/kg/min for 51 hours
  Other Names: GLP-1
  Arms: Active
Drug: Placebo — continuous subcutaneous placebo infusion at a dose of 4.8 pmol/kg/min for 51 hours
  Arms: Placebo

SUMMARY:
GLP-1 is an incretin hormone that simulates insulin secretion and inhibits glucagon secretion in a glucose dependent way. Below normal plasma glucose levels the effects of GLP-1 stop and the risk of hypoglycemia is small. However no results exits on the effects pharmacologically relevant doses of GLP-1 during long-time fasting. There seems to be a risk of hypoglycemia in healthy people after a fasting period when a glucose load is administered. The risk of hypoglycemia when GLP-1 is administered will be evaluated during these two conditions.

DETAILED DESCRIPTION:
GLP-1 is an incretin hormone that simulates insulin secretion and inhibits glucagon secretion dependent on a normal plasma glucose.It also inhibits gastric emptying and has a trophic effect on the pancreatic beta-cells. Below normal plasma glucose levels the effects of GLP-1 stop and the risk of hypoglycemia is small.The counter regulatory response to hypoglycemia has been shown to be preserved during GLP-1 infusion. However no results exits on the effects pharmacologically relevant doses of GLP-1 during long-time fasting. There seems to be a risk of hypoglycemia in healthy people after a fasting period when a glucose load is administered. The risk of hypoglycemia when GLP-1 is administered will be evaluated during these two(48 hours of fasting followed by a glucose-load)conditions in healthy men.

Also the effect on 24 hour blood pressure will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 20-50 years, BMI 20-30 kg/m2, Blood pressure < 140/90 mmHg, caucasian.

Exclusion Criteria:

* Diabetes in relatives, anaemia, any significant disease, smoking.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2005-12; Primary Completion 2006-10 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC)for plasma glucose, insulin, insulin secretion velocity and glucagon for the periods 0-48 hours(day 1-2) and 0-180 min (day 3). And also the lowest plasma glucose during the period 0-180 min day 3 and mean blood pressure | measured every 4 hours for 48 hours (day 1-2) and every 15-30 minutes(day 3)

CONTACTS AND LOCATIONS:
Overall Officials: Ole E. Schmitz, Professor, Principal Investigator — Department of pharmacology, Aarhus university; Birgitte Brock, MD, Study Director — Department of Pharmacology ,University of Aarhus
Locations (1):
- Department of pharmacology, Aarhus university and Medical department M, Aarhus University hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Lerche S, Soendergaard L, Rungby J, Moeller N, Holst JJ, Schmitz OE, Brock B. No increased risk of hypoglycaemic episodes during 48 h of subcutaneous glucagon-like-peptide-1 administration in fasting healthy subjects. Clin Endocrinol (Oxf). 2009 Oct;71(4):500-6. doi: 10.1111/j.1365-2265.2008.03510.x. Epub 2008 Dec 15. PMID 19094067